CLINICAL TRIAL: NCT04479241
Title: A Phase 2, Open-label, Single-arm Study Evaluating the Efficacy, Safety and Tolerability of Lerapolturev (PVSRIPO) and the Immune Checkpoint Inhibitor Pembrolizumab in the Treatment of Patients With Recurrent Glioblastoma
Brief Title: LUMINOS-101: Lerapolturev (PVSRIPO) and Pembrolizumab in Patients With Recurrent Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Istari Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUMINOS-101
Record Dates: First submitted 2020-07-16; First posted 2020-07-21 (Actual); Results first posted 2025-03-25 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-04

CONDITIONS: Glioblastoma; Recurrent Glioblastoma; Supratentorial Glioblastoma; Brain Tumor
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- lerapolturev + pembrolizumab (Experimental): Lerapolturev delivered once intratumorally via convection enhanced delivery. Pembrolizumab given intravenously every 3 weeks.
  Interventions: Biological: lerapolturev; Biological: pembrolizumab

INTERVENTIONS:
Biological: lerapolturev — Lerapolturev (5x10^7 TCID50) delivered intratumorally via convection enhanced delivery (CED).
Biological: pembrolizumab — Pembrolizumab (200 mg IV) given every 3 weeks.

SUMMARY:
This Phase 2 single arm trial in patients with rGBM will characterize the efficacy, safety, tolerability and initial efficacy of lerapolturev intratumoral infusion followed by intravenous pembrolizumab 14 to 28 days later, and every 3 weeks, thereafter.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age.
2. Recurrent supratentorial glioblastoma (GBM) confirmed via prior histology by the site's neuropathologist or designate.

   * Histologically confirmed recurrent glioblastoma (rGBM) within 6 weeks of Lerapolturev infusion will not require a biopsy to confirm active tumor prior to catheter placement
   * Progression of primary glioblastoma or transformation from a lower grade to a higher grade is acceptable for recurrence and as for primary glioblastoma, must be confirmed via prior histology by site pathologist
3. Enhancing lesion ≥1 cm shortest diameter to ≤ 5.5 cm longest diameter in all planes.
4. Before catheter placement based on screening MRI and at the time of catheter placement via CT prior to infusion, neurosurgical investigator must confirm placement of infusion catheter within or through the progressive enhancing tumor is feasible and at a safe distance relative to eloquent brain function, with the tip of the catheter being placed:

   1. Within the enhancing portion or in the vicinity of enhancement of target lesion (ie, infiltrative disease).
   2. ≥ 0.5 cm from ventricles.
   3. ≥ 1 cm deep into the brain.
   4. ≥ 0.5 cm from corpus callosum.
5. First or second relapse supported by MRI or CT scan; relapse is defined as progression following initial/prior therapy(ies).
6. Failed previous first line therapy: maximum surgical resection and radiotherapy (RT) (plus concomitant chemotherapy followed by maintenance chemotherapy if unknown or methylated O6-methylguanine-DNA methyltransferase (MGMT) promoter). Patients who begin but do not complete chemotherapy/RT may still be considered for eligibility at the discretion of Sponsor.
7. Karnofsky Performance Status ≥ 70 at screening and baseline.
8. Undergone prior vaccination against PV and received a boost immunization with trivalent inactivated poliovirus vaccine (IPOL®) at least 1 week, but less than 6 weeks, prior to administration of Lerapolturev. Note: Patients who are unsure of their prior vaccination status/who have not been vaccinated must provide proof of vaccination and/or evidence of anti-PV immunity prior to enrollment, as applicable.
9. Ability to safely discontinue anti-coagulant therapy(ies) prior to biopsy/catheter placement, as required per site/surgical guidelines.
10. Hemoglobin ≥ 9 g/dL prior to biopsy/catheter placement.
11. Platelet count ≥ 100,000/μL (unsupported); ≥ 125,000/ μL (can be supported via platelet transfusion) at biopsy/catheter placement.
12. Absolute Neutrophil Count (ANC) ≥ 1000/μL prior to biopsy/catheter placement.
13. Creatinine ≤ 1.2 x Upper Limit of Normal (ULN) prior to biopsy/catheter placement.
14. Total bilirubin, Alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP) ≤ 2.5 x ULN prior to biopsy/catheter placement.
15. Prothrombin time (PT) and activated Partial Thromboplastin Time (aPTT) ≤ 1.2 x ULN prior to biopsy/catheter placement.
16. If undetectable antitetanus toxin (ATT) Immunoglobulin G (IgG) at screen, Tdap booster vaccine ≥ 1 week prior to biopsy/catheter placement.
17. Patients must be willing and able to understand and provide written informed consent.

Exclusion Criteria:

1. Received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti- CTLA-4 antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways) ≤ 12 weeks prior to lerapolturev infusion (Note: does not apply for patients treated with pembrolizumab under this protocol who are eligible for lerapolturev retreatment). Note: patients who had previously permanently discontinued any anti-PD-1 or PD-L1 therapy due to severe or life-threatening immune-related adverse events are excluded.
2. Excluded are:

   1. Neoplastic lesions in the brainstem, cerebellum, or spinal cord.
   2. Radiological evidence of active/growing multifocal disease: no size increase > 0.5 cm in any direction of any other enhancing non-target lesions present at baseline confirmed via most recent, prior, consecutive MRIs at least 3 months apart.
   3. Tumors with ≥ 1cm of contrast-enhancing tumor component crossing the midline (crossing the corpus callosum).
   4. Extensive subependymal disease: multiple lesions or lesions covering > 50% of subependymal space. Tumor touching subependymal space allowed.
   5. Extensive leptomeningeal disease: multiple lesions or lesions covering > 50% of leptomeninges. Tumor touching leptomeninges allowed.
3. Has received systemic immunosuppressive treatments other than systemic corticosteroids (eg, methotrexate, chloroquine, azathioprine) within six months of Lerapolturev infusion.
4. Requires treatment with high dose systemic corticosteroids, defined as dexamethasone > 4 mg/day or equivalent, within 2 weeks of Lerapolturev infusion.
5. Prior interstitial brachytherapy, implanted chemotherapy, stereotactic radiosurgery or therapeutics delivered by local injection or CED, including Lerapolturev (except for qualifying patients being retreated with Lerapolturev within this trial).
6. Pregnant and/or breast feeding female; patient/female partner of childbearing potential who is unwilling to utilize protocol-defined acceptable form of contraception for duration of study.
7. Impending/life-threatening cerebral herniation syndrome, per neurosurgeon/designate.
8. Severe, active co-morbidity, defined as follows:

   1. Infection requiring IV treatment/unexplained febrile illness (Tmax > 99.5°F/37.5°C)
   2. Known immunosuppressive disease/human immunodeficiency virus infection
   3. Known active hepatitis B or C infection via positive viral DNA or RNA, respectively
   4. Unstable or severe intercurrent medical conditions such as severe heart disease (New York Heart Association Class 3 or 4)
   5. Known lung disease with forced expiratory volume in 1st second of expiration < 50%
   6. Uncontrolled diabetes mellitus (eg, hemoglobin A1C level > 7.0% with treatment)
   7. History of other malignancy requiring active treatment within 2 years of biopsy/catheter placement with the exception of those with a negligible risk of metastasis or death (eg, resected cutaneous basal cell carcinoma, or other cancers with 5-year overall survival (OS) of >90%)
9. Known albumin allergy.
10. Uncontrolled unexplained bleeding and/or hemoptysis within 4 weeks of planned lerapolturev infusion.
11. Inability to undergo brain MRI with and without contrast. History of severe/anaphylactic reaction to gadolinium contrast agent is excluded. Mild allergy (eg, rash) acceptable with prophylactic acetaminophen and diphenhydramine.
12. History of neurological complications due to PV infection.
13. Not recovered from toxic side effects (alopecia acceptable) and/or no current or prior tumor treatments within the following timeframe relative to biopsy/catheter placement:

    1. Chemotherapy or bevacizumab ≤ 4 weeks (except for nitrosourea (6 weeks) or metronomic dosed chemotherapy/targeted therapies such as daily temozolomide, etoposide or cyclophosphamide (1 week)).
    2. Tumor treating fields ≤ 7 days.
    3. RT of brain ≤ 12 weeks, except for progressive disease outside of the radiation field or 2 progressive scans at least 4 weeks apart or histopathologic confirmation.
14. History of agammaglobulinemia.
15. Known hypersensitivity to pembrolizumab, or any components of pembrolizumab.
16. Active autoimmune disease requiring systemic immunomodulatory treatment within the past 12 months; physiologic replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment.
17. History of other malignancy requiring active treatment within 2 years of biopsy/catheter placement with the exception of those with a negligible risk of metastasis or death (eg, resected cutaneous basal cell carcinoma, or other cancers with 5-year OS of >90%)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Franklin, Study Director — Istari Oncology
Locations (10):
- United States (10):
  - University of California San Francisco, San Francisco, California
  - UConn Health, Farmington, Connecticut
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Duke University Medical Center, Durham, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon

RESULTS

PARTICIPANT FLOW:
Groups:
- Lerapolturev + Pembrolizumab: Lerapolturev (5x10^7 TCID50) delivered intratumorally via convection enhanced delivery (CED).
  Pembrolizumab (200 mg IV) given intravenously every 3 weeks.
Period: Overall Study
Arm/Group | Lerapolturev + Pembrolizumab
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lerapolturev + Pembrolizumab
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 22
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 25
Karnofsky Performance Status [Count of Participants; unit: Participants] — KPS is a clinical tool to assess a patient's functional abilities and overall health status. The KPS is a 0-100 point scale where 100 is normal activity with no limitations and 0 is dead. Higher scores indicate a better functional status. A lower score may suggest a poorer prognosis and a greater need for medical care.
  Participants
    80 | 8
    90 | 13
    100 | 4

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Objective response rate (comprised of patients meeting an objective radiographic response or ORR): Patients achieving a complete response (CR) or partial response (PR).
Time Frame: 24 months
Population: No CR or PR were documented; therefore, DOR and DRR cannot be assessed.
Measure: Number; unit: participants
Arm/Group | Lerapolturev + Pembrolizumab
Number analyzed (Participants) | 25
participants | 0

2. Primary Outcome: Frequency and Severity of Treatment-emergent Adverse Events
Description: Count of participants experiencing a treatment-emergent adverse event is reported here. Detailed frequency and severity data are reported in the Adverse Event table.
Time Frame: Up to 30 days after discontinuation of pembrolizumab
Population: patients receiving PVSRIPO and at least one dose of pembrolizumab
Measure: Count of Participants; unit: Participants
Arm/Group | Lerapolturev + Pembrolizumab
Number analyzed (Participants) | 25
Participants | 25

3. Secondary Outcome: Disease Control Rate (DCR)
Description: Proportion of patients achieving stable disease (SD), CR or PR via protocol-specified response criteria
Time Frame: 24 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lerapolturev + Pembrolizumab
Number analyzed (Participants) | 25
percentage of participants | 4 [0 to 14]

4. Secondary Outcome: Survival Assessed by Kaplan-Meier Methods
Description: Overall survival (months) post-lerapolturev infusion estimated by Kaplan-Meier methods.
Time Frame: 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lerapolturev + Pembrolizumab
Number analyzed (Participants) | 25
months | 10.2 [8.9 to 15.9]

5. Primary Outcome: Duration of Response (DOR)
Description: DOR: Time from first ORR observed (once confirmed) until PD first observed (once confirmed) or death; whichever comes first.
Time Frame: 24 months
Population: No CR or PR were documented; therefore, DOR cannot be assessed.
Arm/Group | Lerapolturev + Pembrolizumab
Number analyzed (Participants) | 0

6. Primary Outcome: Durable Radiographic Response (DRR)
Description: DRR: An ORR that persists for ≥ 6 months.
Time Frame: 24 months
Population: No CR or PR were documented; therefore, DRR cannot be assessed.
Arm/Group | Lerapolturev + Pembrolizumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 30 days after the last infusion of pembrolizumab, up to 24 months
Arm/Group | Lerapolturev + Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 25/25
Serious Adverse Events (participants affected / at risk) | 8/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lerapolturev + Pembrolizumab (N=25)
hemiparesis (Nervous system disorders) | 2
brain oedema (Nervous system disorders) | 1
haemorrhage intracranial (Nervous system disorders) | 1
headache (Nervous system disorders) | 1
seizure (Nervous system disorders) | 1
peritumoural oedema (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
pneumonia (Infections and infestations) | 1
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
craniotomy (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lerapolturev + Pembrolizumab (N=25)
headache (Nervous system disorders) | 20
hemiparesis (Nervous system disorders) | 13
seizure (Nervous system disorders) | 9
aphasia (Nervous system disorders) | 4
cognitive disorder (Nervous system disorders) | 4
dizziness (Nervous system disorders) | 4
paraesthesia (Nervous system disorders) | 4
brain oedema (Nervous system disorders) | 3
hemianopia homonymous (Nervous system disorders) | 3
amnesia (Nervous system disorders) | 2
dysarthria (Nervous system disorders) | 2
facial paralysis (Nervous system disorders) | 2
visual field defect (Nervous system disorders) | 2
nausea (Gastrointestinal disorders) | 11
vomiting (Gastrointestinal disorders) | 7
constipation (Gastrointestinal disorders) | 4
diarrhoea (Gastrointestinal disorders) | 4
gastrooesophageal reflux disease (Gastrointestinal disorders) | 4
dysphagia (Gastrointestinal disorders) | 2
fatigue (General disorders) | 14
gait disturbance (General disorders) | 4
pyrexia (General disorders) | 2
lymphocyte count decreased (Investigations) | 3
alanine aminotransferase increased (Investigations) | 2
insomnia (Psychiatric disorders) | 4
agitation (Psychiatric disorders) | 2
confusional state (Psychiatric disorders) | 2
hyperglycaemia (Metabolism and nutrition disorders) | 3
hyponatraemia (Metabolism and nutrition disorders) | 3
decreased appetite (Metabolism and nutrition disorders) | 2
hypoalbuminaemia (Metabolism and nutrition disorders) | 2
hypocalcaemia (Metabolism and nutrition disorders) | 2
arthralgia (Musculoskeletal and connective tissue disorders) | 3
back pain (Musculoskeletal and connective tissue disorders) | 3
myalgia (Musculoskeletal and connective tissue disorders) | 3
flank pain (Musculoskeletal and connective tissue disorders) | 2
peritumoural oedema (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7
epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
cough (Respiratory, thoracic and mediastinal disorders) | 2
photopsia (Eye disorders) | 2
urinary tract infection (Renal and urinary disorders) | 2
rash maculo-papular (Skin and subcutaneous tissue disorders) | 3
dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2
hypertension (Vascular disorders) | 4
anaemia (Blood and lymphatic system disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. The sponsor cannot extend the embargo. The sponsor may request removal of confidential information that does not affect the complete and accurate presentation or interpretation of results.

DOCUMENTS (2):
  • Study Protocol (2021-05-26): https://cdn.clinicaltrials.gov/large-docs/41/NCT04479241/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-23): https://cdn.clinicaltrials.gov/large-docs/41/NCT04479241/SAP_001.pdf